CLINICAL TRIAL: NCT05666973
Title: A Comparative Study on Electrocautery Versus Scalpel for Skin Incision in Inguinal Hernia Repair : A Randomized Controlled Trial
Brief Title: To Compare the Skin Incision Made by the Electrocautery and Scalpel in Inguinal Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Sanjeeb Kumar Jha, Master of Surgery Resident, General Surgery, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SKJha
Record Dates: First submitted 2022-12-15; First posted 2022-12-28 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Post-operative Pain, Acute
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Participants are assigned to study where two groups of treatments Group 1 (Scalpel) and Group 2 (Electrocautery) are given so that Group 1 will receive skin incision only by Scalpel and another group will receive skin incision by Electrocautery for the duration of study.
Who Masked: Participant, Investigator
Masking Description: Patients will be randomly distributed in two groups manually by writing specific numbers that will be concealed in sequentially numbered, opaque sealed envelopes. The envelopes will be opened by an attending nurse not involved in the study just before the procedure. The incision will be given by the attending general surgery resident who will perform the inguinal hernia repair. The assessment of pain and data collection, data analysis will be done by principle investigator who is blinded to procedure. Thus, the patients and investigating and analyzing personal will be blinded to the procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Scalpel (Active Comparator): Skin Incision for inguinal hernia repair will be given by Stainless steel blade no.10.
  Open Mesh Hernioplasty
  Interventions: Procedure: Open Mesh Hernioplasty
- Group 2 : Electrocautery (Experimental): Open Mesh Hernioplasty
  Skin Incision for inguinal hernia repair will be given by following:
  * Cautery machine: Erbe VIO 300 S
  * Cut setting: Cut:30 Coagulate:30
  * Cautery tip (tip pointed)
  * Mode: Monopolar
  Interventions: Procedure: Open Mesh Hernioplasty

INTERVENTIONS:
Procedure: Open Mesh Hernioplasty — * Steps of surgery:
    * Injection Ceftriaxone 50 mg/kg iv stat dose will be given pre-operatively
    * Incision:
  * Incision given over medial 3/5 and 2.5 cms above and parallel to inguinal ligament extending from pubic tubercle upto 1 cm lateral to mid point of inguinal ligament.
    * bleeding controlled by forcep coagulation.
    * Cut the subcutaneous tissues,external oblique aponeurosis opened in layers
    * Nerve Iliohypogastric & ilioinguinal will be preserved (by taking aside from the field)
    * Intra-operative Injection Tramadol(50 mg) and ondansetron(4 mg) iv stat dose given
    * Sac ligated with Polygalactin 2-0 suture.
    * Lichtenstein method of repair
  * Mesh type: large pore polypropylene mesh
  * Mesh size: 3 x 6 inches(7.5 x 15 cms)
  * Mesh Fixation: polypropylene 2-0
    * External oblique closure
    * Skin closure: Ethilon 2 - 0 suture

SUMMARY:
The Groin hernia repair is a commonly performed general surgery procedure in both adults and children with inguinal hernias constituting more than 95% of all groin hernia repairs. Inguinal hernia repair is a commonly performed surgical procedure in our part of the world and is one of the common cause of hospital admission from the emergency or out patient department. Traditionally, surgical skin incisions have been made with surgical scalpel while modern method of making incisions with electrocautery had made it more sharp, precise and less time consuming.

The cases of inguinal hernia are being managed in our center, Tribhuvan University Teaching Hospital. Generally, these patients are seen by the residents and supervised by the faculties in the emergency and in OPD and later if required admitted in the wards. Clinical examination and imaging are done for the diagnosis . Then severity assessment is performed and the management is done accordingly.

The proposed study will be a hospital based comparative study and aims to observe the overview of the surgical management of OPD based day care surgery of inguinal hernia and also to observe whether the surgical incision is being performed with scalpel or electrocautery. The patients fulfilling the inclusion criteria are selected for the study. Sample will be selected by non-probability (convenience) method and study variables will be recorded in proforma. Statistical analysis will be done using SPSS version 23. Results obtained from the study will be reviewed and discussed with published literature.

DETAILED DESCRIPTION:
Inguinal hernia is formed by the protrusion of the peritoneum with its contents through an opening; and the contents - that is, any tissue or organ that protrudes through the neck into the hernia sac. The inguinal hernias are either direct or indirect and both types of hernias protrude above the inguinal ligament.1 Incision is a cut or slit to gain access to underlying structures . Cauterization is a medical term describing burning of body skin to remove or close a part of it. Electrocautery is used increasingly for tissue dissection, although fears of excessive scarring and poor wound healing have curtailed its widespread use for skin incision.2

Traditionally, surgical skin incisions have been made with steel blade. This method of making skin incision is an old method and surgeons have always been in search of some new methods for making surgical skin incisions because incision made by scalpel were supposed to be more bloody, time consuming and more painful.3 Electrocautery which is available in all surgical theaters is less frequently used for skin incisions for the fear of tissue damage, fear of post operative pain and scarring. Recent advances and studies have shown that electrocautery can be used for skin incision without any postoperative complications like wound infection and scarring and less post operative pain.4,5

It has now become an integral and evolving part of surgical practice. However, most surgeons still make skin incision with a scalpel and divide the deeper structures with coagulation diathermy. Modern surgical scalpels are usually made of hardened steel for better sharpness and precision. Basic scalpel design has remained almost the same but there has been a substantial improvement in the electrosurgical instruments.5 Fear of deep burns with diathermy and the resultant scarring continues compared with the scalpel, which produces a clean, incised wound with minimal tissue destruction. Cutting diathermy incision with an electrode delivering pure sinusoidal current allows tissue cleavage by rapid cell vaporization without damage to surrounding areas. This may explain the absence of tissue charring and subsequent healing with minimal scarring. Cutting diathermy can make hemostasis quicker and satisfactory, save the operative time, and can produce an incised wound that heals like the one created by cold scalpel.6,7 Many other studies have been conducted to compare electrocautery skin incision over scalpel skin incision in terms of time taken for incision, postoperative pain and wound healing especially in cases of inguinal hernia surgery, some have reported that the use of diathermy for skin incision during inguinal hernioplasty is as safe as the use of scalpel in terms of wound healing .4

There are other studies which reported that the use of diathermy reduces the use of analgesics requirements in the postoperative period. But still, some studies have reported that the postoperative analgesic requirement are similar in both the techniques and likewise postoperative complications. This study is undertaken to alleviate the fear of using electrocautery for skin incisions in surgical community.

Patients with the provisional diagnosis of inguinal hernia were seen by the residents and supervised by the faculty in the emergency. The severity grading of those patients were done and later admitted in the ward for further management accordingly.

Field Block(Infiltration):

Anesthetic agent:

* Local:

  * Lidoocaine hydrochloride 2% with Adrenaline 1:2,00,000
  * Each ml ;Lidocaine 20mg, Adrenaline 5mcg
  * Maximum safe dose: 7mg/kg (maximum 500mg;25 ml)
* Local

  * Bupivacaine hydrochloride 0.5%
  * Each ml ;Bupivacaine hydrochloride 5 mg
  * Maximum safe dose: 3mg/kg (maximum 225mg;45 ml)
* Local Anesthesia:

  - Field block : With 20 ml Lidocaine 2% and 10 ml Bupivacaine 0.5 % mixed with 20 ml Normal Saline and infiltration in the desired field done.
* Steps of surgery:

  * Injection Ceftriaxone 50 mg/kg iv stat dose will be given pre-operatively
  * Incision:
* medial 3/5 and 2.5 cms above and parallel to inguinal ligament extending from pubic tubercle upto 1 cm lateral to mid point of inguinal ligament.

  * Group 1- Incision with scalpel , bleeding controlled by forcep coagulation.
  * Group 2- Incision with electro cautery needle, hemostasis will be achieved with electrocautery coagulation.
  * Cut the subcutaneous tissues,external oblique aponeurosis opened in layers
  * Nerve Iliohypogastric & ilioinguinal will be preserved (by taking aside from the field)
  * Intra-operative Injection Tramadol(50 mg) and ondansetron(4 mg) iv stat dose given
  * Sac ligated with Polygalactin 2-0 suture.
  * Lichtenstein method of repair
* Mesh type: large pore polypropylene mesh
* Mesh size: 3 x 6 inches(7.5 x 15 cms)
* Mesh Fixation: polypropylene 2-0

  * External oblique closure
  * Skin closure: Ethilon 2 - 0 suture
* Postoperative:

  * Antibiotic:
  * Tab. Cefixime 200 mg PO x BD x 5 days
  * Analgesic :
* Tab Paracetamol 1gm PO x QID x 3 days and SOS
* Tab ketorolac 10 mg PO x SOS
* Tab Pantoprazole 40 mg PO x OD x 5 days The medical records including vital signs, laboratory data, medications and physical examination findings of patients would be reviewed throughout their hospitalization period.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old who are operated with the diagnosis of inguinal hernia.

Exclusion Criteria:

* Patients with recurrent inguinal hernia
* Patients presenting with incarcerated, irreducible and strangulated hernia
* Bilateral Inguinal Hernia
* Patient taking steroids
* Patient with contraindication to NSAIDs such as CKD, Drug hypersensitivity etc
* Patients who do not give written consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
To Compare the incidence of post-operative pain between two groups. | Assessment of Pain will be done • immediately after surgery, 30 minutes , 1 hour • Day 1 to day 5 (Telephone conversation)
  For assessment of pain; visual analog scale will be used in every patients.

SECONDARY OUTCOMES:
To compare the post-operative analgesic dose requirement between the two groups. | Day 1 to Day 5
  For assessment of analgesic dose requirement; will be asked using the telephone conversation.
To Compare the incidence of other complications like SSI, Hematoma, Seroma and Urinary retention between the two groups. | Day 1 to Day 5
  For assessment of other post-operative complications ; patient will be followed up in OPD after telephone conversation.

CONTACTS AND LOCATIONS:
Overall Officials: Yogendra Pd Singh, MBBS,MS, Study Chair — Tribhuvan University Teaching Hospital, Institute Of Medicine.

IPD SHARING:
Plan to Share IPD: No